CLINICAL TRIAL: NCT05536687
Title: VALIDITY AND RELIABILITY OF THE 6-MINUTES WALKING TEST EVALUATED BY FEETME® INSOLES
Acronym: ValiFeet6
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: minimum of participants reached and lack of ressources for recruitment
Sponsor: FeetMe (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ValiFeet6
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Healthy
Keywords: Healthy; 6MWT; Real-world; insoles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy (Other)
  Interventions: Device: FeetMe

INTERVENTIONS:
Device: FeetMe — Healthy volunteers will wear the insoles at 2 visits in hospitals (D0 and D8) and 2 visits at home (D1 and D7). The visits at the hospital will be composed of 3 tests of 6 min. in various conditions in a hospital environment :
  * In degraded conditions, i.e. a 10m corridor, evaluated simultaneously by the FeetMe® system and an evaluator
  * In degraded condition, a 10m corridor, evaluated simultaneously by the FeetMe® system and an odometer and evaluator
  * Under the conditions recommended for the 6-minute test (ref), i.e. a 30m corridor, evaluated simultaneously by the FeetMe® system and the evaluator A rest time of 15 min minimum will be respected between each test. The visits at home will be composed of a 6-minute test at home or outdoors (quiet place, flat, hard surface, few or no passages, ideally no obstacles, covered if weather conditions are not suitable) with a 10-meter track that you can define simply with equipment provided by the promoter.

SUMMARY:
Currently, the guidelines for performing the 6MWT established by the American Thoracic Society and the European Respiratory Society (ATS/ERS) recommend the use of an indoor or outdoor corridor with a 30 m flat surface (6MWT30) for patients with respiratory diseases, which is also a recommendation for healthy adults. However, not all hospitals, nursing homes or clinics have a corridor of sufficient length to properly perform the 6MWT. A simple way to make the test available to more health care professionals would be to reduce the length of the hallway.

In times when access to the hospital is difficult, the ability to assess functional abilities at a distance becomes essential. Today, this is becoming possible with tools such as connected watches, accelerometers, connected shoes and insoles. They give access to a quantitative analysis of walking without necessarily requiring large spaces, specialized personnel or even being in a hospital environment. The FeetMe® Evaluation device consists of connected insoles as well as a mobile application allowing the evaluation of standard clinical walking tests.

This device allows a better understanding of patients' walking and is transposable in real life.

The objective of the present study is to demonstrate the validity and reliability of the measurement of the distance walked during a 6-minute test with connected insoles in standard conditions (6MW30), degraded conditions (6MW10) in a clinic and at home in a healthy population divided into age subgroups.

In addition, this study will investigate whether there is a relationship between 6 minutes of uncontrolled walking from real-life walking data and a standard 6-minute test.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 80 years old

  * Able to use a laptop
  * Able to walk 100 meters without any aid
  * Accustomed to using a smartphone

Exclusion Criteria:

* Surgery with the possibility of impacting gait in the previous 3 months having had an impact on gait: orthopedic surgery, trauma of the lower limbs and spine, gynecological or urological surgery, brain and spinal cord surgery • Chronic disease affecting walking: Rheumatological, orthopedic, painful, neurological pathology.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Reliability of the test-retest for the distance during a 6MWT | 10 days
  Compare the reliability of the test-retest for the distance evaluated by the FeetMe® solution during a 6MWT10 performed at home (6MWT10-Home) compared to a 6MWT10 performed in a hospital setting (6MWT10-Hospital).

CONTACTS AND LOCATIONS:
Locations (1):
- Ch Delafontaine, Saint-Denis, France

IPD SHARING:
Plan to Share IPD: Undecided